CLINICAL TRIAL: NCT02561156
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Safety, Tolerability and Pharmacokinetic Study of Escalating Single and Multiple Doses of TAK-653 in Healthy Subjects
Brief Title: TAK-653 Escalating Single and Multiple Dose Study in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: TAK-653-1001; 2015-002268-17 (EudraCT Number); U1111-1170-0519 (Registry Identifier: WHO); 15/SS/0117 (Registry Identifier: NRES)
Record Dates: First submitted 2015-09-09; First posted 2015-09-25 (Estimated); Results first posted 2019-02-08 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Depressive Disorder
Keywords: Drug therapy
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (13):
- Part 1 Cohort 1: TAK-653 0.3 mg (Experimental): TAK-653 0.3 milligram (mg), tablet, orally, once on Day 1 or TAK-653 placebo-matching tablet, orally, once on Day 1. TAK-653 or placebo will be administered after an overnight fast of approximately at least 10 hours.
  Interventions: Drug: TAK-653 Placebo; Drug: TAK-653
- Part 1 Cohort 2: TAK-653 1.0 mg (Experimental): TAK-653 1.0 mg, tablet, orally, once on Day 1 or TAK-653 placebo-matching tablet, orally, once on Day 1. TAK-653 or placebo will be administered after an overnight fast of approximately at least 10 hours.
  Interventions: Drug: TAK-653 Placebo; Drug: TAK-653
- Part 1 Cohort 3: TAK-653 3.0 mg (Experimental): TAK-653 3.0 mg, tablet, orally, once on Day 1 or TAK-653 placebo-matching tablet, orally, once on Day 1. TAK-653 or placebo will be administered after an overnight fast of approximately at least 10 hours.
  Interventions: Drug: TAK-653 Placebo; Drug: TAK-653
- Part 1 Cohort 4: TAK-653 5.0 mg (Experimental): TAK-653 5.0 mg, tablet, orally, once on Day 1 or TAK-653 placebo-matching tablet, orally, once on Day 1. TAK-653 or placebo will be administered after an overnight fast of approximately at least 10 hours.
  Interventions: Drug: TAK-653 Placebo; Drug: TAK-653
- Part 1 Cohort 5: TAK-653 9.0 mg (Experimental): TAK-653 9.0 mg, tablet, orally, once on Day 1 or TAK-653 placebo-matching tablet, orally, once on Day 1. TAK-653 or placebo will be administered after an overnight fast of approximately at least 10 hours.
  Interventions: Drug: TAK-653 Placebo; Drug: TAK-653
- Part 1 Cohort 6: TAK- 653 18 mg (Experimental): TAK-653 18 mg, tablet, orally, once on Day 1 or TAK-653 placebo-matching tablet, orally, once on Day 1. TAK-653 or placebo will be administered after an overnight fast of approximately at least 10 hours. Dose escalation to be decided (TBD) based on safety, tolerability, and available PK and pharmacodynamics (PD) data from previous cohorts.
  Interventions: Drug: TAK-653 Placebo; Drug: TAK-653
- Part 1 Additional Cohorts: TAK- 653 Placebo (Experimental): TAK-653 placebo-matching tablet, orally, once on Day 1. TAK-653 or placebo will be administered after an overnight fast of approximately at least 10 hours. Dose escalation TBD based on safety, tolerability, and available PK and PD data from previous cohorts.
  Interventions: Drug: TAK-653 Placebo; Drug: TAK-653
- Part 2 Cohort 1: TAK-653 0.3 mg (Experimental): TAK-653 0.3 mg, tablet, orally, once on Day 1, and once daily (QD) from Days 6 to 18 or placebo-matching tablet, orally, once on Day 1 and QD from Days 6 to 18.
  Interventions: Drug: TAK-653 Placebo; Drug: TAK-653
- Part 2 Cohort 2: TAK-653 1.0 mg (Experimental): TAK-653 1.0 mg, tablet, orally, once on Day 1, and QD from Days 6 to 18 or placebo-matching tablet, orally, once on Day 1 and QD from Days 6 to 18.
  Interventions: Drug: TAK-653 Placebo; Drug: TAK-653
- Part 2 Cohort 3: TAK-653 3.0 mg (Experimental): TAK-653 3.0 mg, tablet, orally, once on Day 1, and QD from Days 6 to 18 or placebo-matching tablet, orally, once on Day 1 and QD from Days 6 to 18.
  Interventions: Drug: TAK-653 Placebo; Drug: TAK-653
- Part 2 Cohort 4: TAK-653 6 mg (Experimental): TAK-653 6 mg, tablet, orally, once on Day 1, and QD from Days 6 to 18 or placebo-matching tablet, orally, once on Day 1 and QD from Days 6 to 18. Dose escalation TBD based on safety, tolerability, and available PK and PD data from previous cohorts.
  Interventions: Drug: TAK-653 Placebo; Drug: TAK-653
- Part 2 Cohort 5: TAK-653 9 mg (Experimental): TAK-653 9 mg, tablet, orally, once on Day 1, and QD from Days 6 to 18 or placebo-matching tablet, orally, once on Day 1 and QD from Days 6 to 18. Dose escalation TBD based on safety, tolerability, and available PK and PD data from previous cohorts.
  Interventions: Drug: TAK-653 Placebo; Drug: TAK-653
- Part 2 Additional Cohorts: TAK-653 Placebo (Experimental): TAK-653 placebo-matching tablet, orally, once on Day 1 and QD from Days 6 to 18. Dose escalation TBD based on safety, tolerability, and available PK and PD data from previous cohorts.
  Interventions: Drug: TAK-653 Placebo; Drug: TAK-653

INTERVENTIONS:
Drug: TAK-653 Placebo — TAK-653 placebo-matching tablets.
Drug: TAK-653 — TAK-653 tablets.

SUMMARY:
The purpose of this study is to assess the safety, tolerability and pharmacokinetics (PK) of TAK-653 when administered as single and multiple oral doses at escalating dose levels in healthy participants.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-653. TAK-653 is being tested to treat people who have depression. This study will look at the tolerability and PK of TAK-653 in healthy participants.

The study may enroll up to 112 participants and each cohort will enroll 8 participants. This study consists of 2 parts: Part 1- single rising dose (SRD) consisting of at least 6 cohorts and Part 2- single rising dose and multiple rising dose (SRD/MRD) consisting of at least 5 cohorts. Additional cohorts may be added depending on the emerging safety and PK data. Participants will be randomly assigned (by chance, like flipping a coin) within each cohort to receive TAK-653 or placebo which will remain undisclosed to the participants and study doctor during the study (unless there is an urgent medical need). Participants enrolled in Cohort 1 to 5 of Part 1 will receive TAK-653 0.3 mg, 1.0 mg, 3.0 mg, 5.0 mg and 9.0 mg or TAK-653 placebo-matching tablet. Subsequent dose escalation in Part-1, from Cohort 6 onward will occur after the full availability of safety, tolerability, PK, and PD data from preceding cohorts. Participants in Part-2 Cohorts 1 to 3 will receive TAK-653 0.3 mg, 1.0 mg and 3.0 mg respectively. Dose for Part 2, from Cohort 4 onward will be based on review of safety, tolerability, and available PK and PD data from previous cohorts. All participants will be asked to take the drug at the same time each day on Day 1 for Part 1 and Day 1 and Days 6 to 18 in Part 2.

This single-center trial will be conducted in the United Kingdom. The overall time to participate in this study is approximately 14 days for Part 1 and 31 days for Part 2. Participants will be admitted to the clinic for 6 days in Part 1 and 22 days in Part 2. Participants will be followed up 14 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Is capable of understanding and complying with protocol requirements.
2. Signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures including requesting that a participant fasts for any laboratory evaluations.
3. Weighs at least 45 kilogram (kg) and has a body mass index (BMI) between 18.0 and 30.0 kilogram per square meter (kg/m^2), inclusive at Screening.
4. Male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 90 days after 5 half-lives have elapsed since last dose of study drug. This should be interpreted as 90 days from the Follow-up Call/Visit unless data indicates otherwise.
5. Female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to routinely use highly effective contraception with low user dependency from signing of informed consent, throughout the duration of the study, and for 30 days after 5 half-lives have elapsed since the last dose of study drug. This should be interpreted as 30 days from the Follow-up Call/Visit unless data indicates otherwise.

Exclusion Criteria:

1. Has received any investigational compound within 90 days prior to the first dose of study drug.
2. Is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in the conduct of this study (example, spouse, parent, child, sibling) or may consent under duress.
3. Has any clinically significant illness, such as cardiovascular, neurologic, pulmonary, hepatic, renal, metabolic, gastrointestinal, urologic, immunologic, endocrine, or psychiatric disease or disorder, or other abnormality, which may affect safety, increase risk of seizure or lower the seizure threshold, or potentially confound the study results. It is the responsibility of the investigator to assess the clinical significance; however, consultation with the Takeda Medical Monitor may be warranted.
4. Has a known hypersensitivity to any component of the formulation of TAK-653.
5. Has taken any excluded medication, supplements, or food products during the time periods.
6. Is pregnant or lactating or intending to become pregnant before, during, or within 30 days after 5 half-lives have elapsed since the last dose of study drug (30 days from the Follow-up Call/Visit unless available data indicates otherwise); or intending to donate ova during such time period.
7. If male, intends to donate sperm during the course of this study or within 90 days after 5 half-lives have elapsed since the last dose of study drug. This should be interpreted as 90 days from the Follow-up Call/Visit unless data indicates otherwise.
8. Has had previous episodes of seizures or convulsion (lifetime), including absence seizure and febrile convulsion.
9. Participant or any immediate family member has a history of epilepsy (including febrile convulsions).
10. Has a history of neurological abnormalities including abnormal EEG at screening or brain injury including traumatic injury, perinatal cerebropathy and postnatal brain damage, blood-brain barrier abnormality, and angioma cavernous.
11. Has a history of cerebral arteriosclerosis.
12. Has a condition that can potentially reduce drug clearance (example, renal or hepatic insufficiency).
13. Has current or recent (within 6 months) gastrointestinal disease that would be expected to influence the absorption of drugs (that is, a history of malabsorption, any surgical intervention known to impact absorption [example, bariatric surgery or bowel resection], esophageal reflux, peptic ulcer disease, erosive esophagitis, or frequent [more than once per week] occurrence of heartburn).
14. Has a history of cancer, except basal cell carcinoma which has been in remission for at least 5 years prior to Check-in (Day 1).
15. Has a positive test result for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, or a known history of human immunodeficiency virus (HIV) infection at Screening.
16. Has poor peripheral venous access.
17. Has a positive urine/blood result for drugs of abuse (defined as any illicit drug use) at Screening or Check-in (Day -1).
18. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 1 year prior to Screening or is unwilling to agree to abstain from alcohol and drugs throughout the study.
19. Has used nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patch, or nicotine gum) within 28 days prior to Check-in Day -1. Cotinine test is positive at Screening or Check-in (Day -1).
20. Has donated or lost 450 milliliter (mL) or more of his or her blood volume (including plasmapheresis), or had a transfusion of any blood product within 90 days prior to first dose of study drug.
21. Has a Screening or Check-in (Day -1) abnormal (clinically significant [CS]) ECG. Entry of any participant with an abnormal (not clinically significant [NCS]) ECG must be approved, and documented by signature of the principal investigator or medically qualified subinvestigator. In the case of a QT interval corrected using Fridericia's formula (QTcF) interval greater than (>) 450 millisecond (msec) or >480 msec (participants with Bundle Branch Block) or PR outside the range of 120 to 220 msec, assessment may be repeated once for eligibility determination at the Screening Visit and/or Check-in (Day -1) Visit.
22. Has a supine blood pressure outside the ranges of greater than or equal to (>=) 90 to less than or equal to (<=)140 millimeter of mercury (mmHg) for systolic and >= 50 to <= 90 mm Hg for diastolic. If out of range, assessment may be repeated once for eligibility determination at the Screening Visit and/or Check-in (Day -1).
23. Has a resting heart rate outside the range of 50 to 90 bpm (not on ECGs). If out of range, the assessment may be repeated once for eligibility determination at the Screening Visit and/or Check-in (Day -1).
24. Has abnormal Screening or Check-in (Day -1) laboratory values that suggest a clinically significant underlying disease or participant has the following lab abnormalities: Alanine transaminase (ALT) and/or Aspartate aminotransferase (AST) >1.5 upper limit of normal (ULN).
25. Has a risk of suicide per the C-SSRS (a score of 4 or 5 on ideation or any suicidal behavior) or according to the investigator's clinical judgment, has made a suicide attempt in the previous 6 months, or has a history of deliberate self-harm in the past 6 months.

Additional exclusion criteria for CSF collection in Cohort 3 in Part 2:

1. Has had CSF collected within 6 months prior to Check-in (Day -1).
2. Has a known hypersensitivity to the anesthetic or its derivatives used during CSF collection or any medication used to prepare the area of lumbar puncture.
3. Has any skin condition, abnormality of the lumbar spine, medical or surgical condition that would preclude lumbar puncture (example, coagulopathy, local or systemic infection, left ventricular outflow obstruction, aortic stenosis, raised intracranial pressure, previous back surgery).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2015-08-26 (Actual); Primary Completion 2017-09-11 (Actual); Study Completion 2017-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (1):
- Hammersmith Medicines Research, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available after applicable marketing approvals and commercial availability have been received, an opportunity for the primary publication of the research has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com/Approach for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in United Kingdom from 26 August 2015 to 23 September 2017.
Pre-assignment Details: Healthy participants were enrolled in this 2 part study to receive TAK-653 as: single rising (SRD) dose of 0.3 milligram (mg), 1 mg, 3 mg , 5 mg, 9 mg or 18 mg in Part 1, and SRD/multiple rising dose (MRD) of 0.3 mg, 1 mg, 3 mg, 6 mg or 9 mg in Part 2.
Groups:
- Part 1 Cohorts 1-6: Pooled Placebo: TAK-653 placebo-matching tablet, orally, once under fasted conditions on Day 1.
- Part 1 Cohort 1: TAK-653 0.3 mg: TAK-653 0.3 mg, tablet, orally, once under fasted conditions on Day 1.
- Part 1 Cohort 2: TAK-653 1 mg: TAK-653 1 mg, tablet, orally, once under fasted conditions on Day 1.
- Part 1 Cohort 3: TAK-653 3 mg+TAK-653 3mg: TAK-653 3 mg, tablet, orally, once, under fasted condition on Day 1 of Period 1 and TAK-653 3 mg, tablet, orally, once, under fed condition on Day 1 of Period 2.
- Part 1 Cohort 4: TAK-653 5 mg: TAK-653 5 mg, tablet, orally, once under fasted conditions on Day 1.
- Part 1 Cohort 5: TAK-653 9 mg: TAK-653 9 mg, tablet, orally, once under fasted conditions on Day 1.
- Part 1 Cohort 6: TAK-653 18 mg: TAK-653 18 mg, tablet, orally, once under fasted conditions on Day 1.
- Part 2 Cohorts 1-5: Pooled Placebo: TAK-653 placebo-matching tablet, orally, once under fasted conditions on Day 1 and Days 6-18.
- Part 2 Cohort 1: TAK-653 0.3 mg: TAK-653 0.3 mg, tablet, orally, once under fasted conditions on Day 1 and Days 6-18.
- Part 2 Cohort 2: TAK-653 1 mg: TAK-653 1 mg, tablet, orally, once under fasted conditions on Day 1 and Days 6-18.
- Part 2 Cohort 3: TAK-653 3 mg: TAK-653 3 mg, tablet, orally, once under fasted conditions on Day 1 and Days 6-18.
- Part 2 Cohort 4: TAK-653 6 mg: TAK-653 6 mg, tablet, orally, once under fasted conditions on Day 1 and Days 6-18.
- Part 2 Cohort 5: TAK-653 9 mg: TAK-653 9 mg, tablet, orally, once under fasted conditions on Day 1 and Days 6-18.
Period: Part 1
Arm/Group | Part 1 Cohorts 1-6: Pooled Placebo | Part 1 Cohort 1: TAK-653 0.3 mg | Part 1 Cohort 2: TAK-653 1 mg | Part 1 Cohort 3: TAK-653 3 mg+TAK-653 3mg | Part 1 Cohort 4: TAK-653 5 mg | Part 1 Cohort 5: TAK-653 9 mg | Part 1 Cohort 6: TAK-653 18 mg | Part 2 Cohorts 1-5: Pooled Placebo | Part 2 Cohort 1: TAK-653 0.3 mg | Part 2 Cohort 2: TAK-653 1 mg | Part 2 Cohort 3: TAK-653 3 mg | Part 2 Cohort 4: TAK-653 6 mg | Part 2 Cohort 5: TAK-653 9 mg
Started | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2
Arm/Group | Part 1 Cohorts 1-6: Pooled Placebo | Part 1 Cohort 1: TAK-653 0.3 mg | Part 1 Cohort 2: TAK-653 1 mg | Part 1 Cohort 3: TAK-653 3 mg+TAK-653 3mg | Part 1 Cohort 4: TAK-653 5 mg | Part 1 Cohort 5: TAK-653 9 mg | Part 1 Cohort 6: TAK-653 18 mg | Part 2 Cohorts 1-5: Pooled Placebo | Part 2 Cohort 1: TAK-653 0.3 mg | Part 2 Cohort 2: TAK-653 1 mg | Part 2 Cohort 3: TAK-653 3 mg | Part 2 Cohort 4: TAK-653 6 mg | Part 2 Cohort 5: TAK-653 9 mg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 6 | 6 | 6 | 6 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 6 | 6 | 6 | 5 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 Cohorts 1-6: Pooled Placebo | Part 1 Cohort 1: TAK-653 0.3 mg | Part 1 Cohort 2: TAK-653 1 mg | Part 1 Cohort 3: TAK-653 3 mg+TAK-653 3mg | Part 1 Cohort 4: TAK-653 5 mg | Part 1 Cohort 5: TAK-653 9 mg | Part 1 Cohort 6: TAK-653 18 mg | Part 2 Cohorts 1-5: Pooled Placebo | Part 2 Cohort 1: TAK-653 0.3 mg | Part 2 Cohort 2: TAK-653 1 mg | Part 2 Cohort 3: TAK-653 3 mg | Part 2 Cohort 4: TAK-653 6 mg | Part 2 Cohort 5: TAK-653 9 mg | Total
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 10 | 6 | 6 | 6 | 6 | 6 | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 10 | 6 | 6 | 6 | 6 | 6 | 88
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
  Male | 10 | 5 | 5 | 6 | 6 | 6 | 6 | 10 | 6 | 6 | 6 | 6 | 6 | 84
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 3
  Not Hispanic or Latino | 12 | 6 | 5 | 6 | 6 | 6 | 5 | 10 | 6 | 6 | 6 | 5 | 6 | 85
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 8
  White | 8 | 6 | 4 | 6 | 6 | 4 | 5 | 7 | 4 | 4 | 5 | 6 | 4 | 69
  More than one race | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 10 | 6 | 6 | 6 | 6 | 6 | 88
Smoking Classification [Count of Participants; unit: Participants]
  Never smoked | 10 | 4 | 5 | 4 | 4 | 4 | 4 | 6 | 4 | 4 | 4 | 5 | 4 | 62
  Ex-smoker | 2 | 2 | 1 | 2 | 2 | 2 | 2 | 4 | 2 | 2 | 2 | 1 | 2 | 26
Female Reproductive Status [Count of Participants; unit: Participants] — Population: Female reproductive status was only assessed in females.
  Participants
    number analyzed (Participants) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
    Surgically sterile | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Female of childbearing potential | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Caffeine Consumption [Count of Participants; unit: Participants]
  Had caffeine consumption | 8 | 6 | 3 | 4 | 5 | 6 | 5 | 9 | 4 | 4 | 4 | 4 | 4 | 66
  Had no caffeine consumption | 4 | 0 | 3 | 2 | 1 | 0 | 1 | 1 | 2 | 2 | 2 | 2 | 2 | 22

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Percentage of Participants Who Experience at Least One Treatment Emergent Adverse Event (TEAE)
Time Frame: Baseline up to Day 14
Population: The safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 Cohorts 1-6: Pooled Placebo | Part 1 Cohort 1: TAK-653 0.3 mg | Part 1 Cohort 2: TAK-653 1 mg | Part 1 Cohort 3: TAK-653 3 mg+TAK-653 3mg | Part 1 Cohort 4: TAK-653 5 mg | Part 1 Cohort 5: TAK-653 9 mg | Part 1 Cohort 6: TAK-653 18 mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
percentage of participants | 41.7 | 66.7 | 66.7 | 50.0 | 83.3 | 33.3 | 33.3

2. Primary Outcome: Part 2: Percentage of Participants Who Experience at Least One TEAE
Time Frame: Baseline up to Day 31
Population: The safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 2 Cohorts 1-5: Pooled Placebo | Part 2 Cohort 1: TAK-653 0.3 mg | Part 2 Cohort 2: TAK-653 1 mg | Part 2 Cohort 3: TAK-653 3 mg | Part 2 Cohort 4: TAK-653 6 mg | Part 2 Cohort 5: TAK-653 9 mg
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
percentage of participants | 50.0 | 50.0 | 50.0 | 100.0 | 33.3 | 50.0

3. Primary Outcome: Part 1: Percentage of Participants Who Discontinued the Treatment Due to an Adverse Event (AE)
Time Frame: Baseline up to Day 14
Population: The safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 Cohorts 1-6: Pooled Placebo | Part 1 Cohort 1: TAK-653 0.3 mg | Part 1 Cohort 2: TAK-653 1 mg | Part 1 Cohort 3: TAK-653 3 mg+TAK-653 3mg | Part 1 Cohort 4: TAK-653 5 mg | Part 1 Cohort 5: TAK-653 9 mg | Part 1 Cohort 6: TAK-653 18 mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Part 2: Percentage of Participants Who Discontinued the Treatment Due to an AE
Time Frame: Baseline up to Day 31
Population: The safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 2 Cohorts 1-5: Pooled Placebo | Part 2 Cohort 1: TAK-653 0.3 mg | Part 2 Cohort 2: TAK-653 1 mg | Part 2 Cohort 3: TAK-653 3 mg | Part 2 Cohort 4: TAK-653 6 mg | Part 2 Cohort 5: TAK-653 9 mg
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
percentage of participants | 0 | 0 | 0 | 0 | 16.7 | 0

5. Primary Outcome: Part 1: Percentage of Participants Who Meet the Markedly Abnormal Criteria for Safety Laboratory Tests at Least Once Postdose
Time Frame: Cohort 1-5: Baseline up to Day 7; Cohort 6: Baseline up to Day 8
Population: The safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 Cohorts 1-6: Pooled Placebo | Part 1 Cohort 1: TAK-653 0.3 mg | Part 1 Cohort 2: TAK-653 1 mg | Part 1 Cohort 3: TAK-653 3 mg+TAK-653 3mg | Part 1 Cohort 4: TAK-653 5 mg | Part 1 Cohort 5: TAK-653 9 mg | Part 1 Cohort 6: TAK-653 18 mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
percentage of participants | 0 | 16.7 | 0 | 16.7 | 0 | 0 | 0

6. Primary Outcome: Part 2: Percentage of Participants Who Meet the Markedly Abnormal Criteria for Safety Laboratory Tests at Least Once Postdose
Time Frame: Baseline up to Day 8
Population: The safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 2 Cohorts 1-5: Pooled Placebo | Part 2 Cohort 1: TAK-653 0.3 mg | Part 2 Cohort 2: TAK-653 1 mg | Part 2 Cohort 3: TAK-653 3 mg | Part 2 Cohort 4: TAK-653 6 mg | Part 2 Cohort 5: TAK-653 9 mg
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
percentage of participants | 0 | 33.3 | 0 | 0 | 0 | 16.7

7. Primary Outcome: Part 1: Percentage of Participants Who Meet the Markedly Abnormal Criteria for Vital Sign Measurements at Least Once Postdose
Time Frame: Cohort 1-5: Baseline up to Day 7; Cohort 6: Baseline up to Day 8
Population: The safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 Cohorts 1-6: Pooled Placebo | Part 1 Cohort 1: TAK-653 0.3 mg | Part 1 Cohort 2: TAK-653 1 mg | Part 1 Cohort 3: TAK-653 3 mg+TAK-653 3mg | Part 1 Cohort 4: TAK-653 5 mg | Part 1 Cohort 5: TAK-653 9 mg | Part 1 Cohort 6: TAK-653 18 mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
percentage of participants | 75.0 | 50.0 | 100.0 | 66.7 | 83.3 | 83.3 | 66.7

8. Primary Outcome: Part 2: Percentage of Participants Who Meet the Markedly Abnormal Criteria for Vital Sign Measurements at Least Once Postdose
Time Frame: Baseline up to Day 21
Population: The safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 2 Cohorts 1-5: Pooled Placebo | Part 2 Cohort 1: TAK-653 0.3 mg | Part 2 Cohort 2: TAK-653 1 mg | Part 2 Cohort 3: TAK-653 3 mg | Part 2 Cohort 4: TAK-653 6 mg | Part 2 Cohort 5: TAK-653 9 mg
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
percentage of participants | 90.0 | 100.0 | 100.0 | 100.0 | 83.3 | 83.3

9. Primary Outcome: Part 1: Percentage of Participants Who Meet the Markedly Abnormal Criteria for Safety Electrocardiogram (ECG) at Least Once Postdose
Time Frame: Cohort 1-5: Baseline up to Day 7; Cohort 6: Baseline up to Day 8
Population: The safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 Cohorts 1-6: Pooled Placebo | Part 1 Cohort 1: TAK-653 0.3 mg | Part 1 Cohort 2: TAK-653 1 mg | Part 1 Cohort 3: TAK-653 3 mg+TAK-653 3mg | Part 1 Cohort 4: TAK-653 5 mg | Part 1 Cohort 5: TAK-653 9 mg | Part 1 Cohort 6: TAK-653 18 mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
percentage of participants | 66.7 | 33.3 | 33.3 | 50.0 | 0 | 33.3 | 50

10. Primary Outcome: Part 2: Percentage of Participants Who Meet the Markedly Abnormal Criteria for Safety ECG at Least Once Postdose
Time Frame: Baseline up to Day 8
Population: The safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 2 Cohorts 1-5: Pooled Placebo | Part 2 Cohort 1: TAK-653 0.3 mg | Part 2 Cohort 2: TAK-653 1 mg | Part 2 Cohort 3: TAK-653 3 mg | Part 2 Cohort 4: TAK-653 6 mg | Part 2 Cohort 5: TAK-653 9 mg
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
percentage of participants | 40.0 | 50.0 | 50.0 | 16.7 | 50.0 | 16.7

11. Primary Outcome: Part 1: Percentage of Participants Who Experience Clinically Significant Abnormal Changes in Safety Electroencephalogram (EEG) Measurements at Least Once Postdose
Time Frame: Cohort 1-5: Baseline up to Day 7; Cohort 6: Baseline up to Day 8
Population: The safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 Cohorts 1-6: Pooled Placebo | Part 1 Cohort 1: TAK-653 0.3 mg | Part 1 Cohort 2: TAK-653 1 mg | Part 1 Cohort 3: TAK-653 3 mg+TAK-653 3mg | Part 1 Cohort 4: TAK-653 5 mg | Part 1 Cohort 5: TAK-653 9 mg | Part 1 Cohort 6: TAK-653 18 mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Primary Outcome: Part 2: Percentage of Participants Who Experience Clinically Significant Abnormal Changes in Safety EEG Measurements at Least Once Postdose
Time Frame: Baseline up to Day 18
Population: The safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 2 Cohorts 1-5: Pooled Placebo | Part 2 Cohort 1: TAK-653 0.3 mg | Part 2 Cohort 2: TAK-653 1 mg | Part 2 Cohort 3: TAK-653 3 mg | Part 2 Cohort 4: TAK-653 6 mg | Part 2 Cohort 5: TAK-653 9 mg
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
percentage of participants | 0 | 0 | 0 | 0 | 0 | 0

13. Primary Outcome: Part 1: Number of Participants With Treatment-emergent Suicidal Ideation or Suicidal Behavior as Measured Using Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: Treatment-emergent suicidal ideation or behavior compared to baseline will be measured by an increase in suicidal ideation category (1-5 on the C-SSRS) or suicidal behavior category (6-10 on the C-SSRS) during treatment from the maximum suicidal ideation/behavior category at baseline, or any suicidal ideation/behavior during treatment if there is none at baseline. C-SSRS is used to assess whether participant experienced suicidal ideation (1: wish to be dead; 2: non-specific active suicidal thoughts; 3: active suicidal ideation with any methods (not plan) without intent to act; 4: active suicidal ideation with some intent to act, without specific plan; 5: active suicidal ideation with specific plan and intent) and suicidal behavior (6: actual attempt; 7: interrupted attempt; 8: aborted attempt; 9: preparatory acts or behavior; 10: suicidal behavior).
Time Frame: Cohort 1-5: Baseline up to Day 7; Cohort 6: Baseline up to Day 8
Population: The safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Part 1 Cohorts 1-6: Pooled Placebo | Part 1 Cohort 1: TAK-653 0.3 mg | Part 1 Cohort 2: TAK-653 1 mg | Part 1 Cohort 3: TAK-653 3 mg+TAK-653 3mg | Part 1 Cohort 4: TAK-653 5 mg | Part 1 Cohort 5: TAK-653 9 mg | Part 1 Cohort 6: TAK-653 18 mg
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-653 on Day 1
Time Frame: Part 1 Cohort 1-5: Day 1 pre-dose and at multiple timepoints (up to 144 hours) post-dose; Part 1 Cohort 6: Day 1 pre-dose and at multiple timepoints (up to 168 hours) post-dose; Part 2: Day 1 pre-dose and at multiple timepoints (up to 120 hours) post-dose
Population: The pharmacokinetics (PK) analysis set included all participants who received study drug and had at least 1 measurable plasma concentration or amount of drug in urine.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part 1 Cohort 1: TAK-653 0.3 mg | Part 1 Cohort 2: TAK-653 1 mg | Part 1 Cohort 3: TAK-653 3 mg+TAK-653 3mg | Part 1 Cohort 4: TAK-653 5 mg | Part 1 Cohort 5: TAK-653 9 mg | Part 1 Cohort 6: TAK-653 18 mg | Part 2 Cohort 1: TAK-653 0.3 mg | Part 2 Cohort 2: TAK-653 1 mg | Part 2 Cohort 3: TAK-653 3 mg | Part 2 Cohort 4: TAK-653 6 mg | Part 2 Cohort 5: TAK-653 9 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
nanogram per milliliter (ng/mL) | 3.5985 (14) | 10.2220 (15) | 26.9733 (10) | 44.9430 (13) | 68.8039 (16) | 123.6462 (21) | 2.8630 (23) | 7.7786 (12) | 28.0546 (23) | 41.0028 (24) | 76.0656 (27)

15. Secondary Outcome: Part 2: Cmax: Maximum Observed Plasma Concentration for TAK-653 on Day 6
Time Frame: Day 6 pre-dose at multiple timepoints (up to 24 hours) post dose
Population: The PK analysis set included all participants who received study drug and had at least 1 measurable plasma concentration or amount of drug in urine.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 2 Cohort 1: TAK-653 0.3 mg | Part 2 Cohort 2: TAK-653 1 mg | Part 2 Cohort 3: TAK-653 3 mg | Part 2 Cohort 4: TAK-653 6 mg | Part 2 Cohort 5: TAK-653 9 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
ng/mL | 3.0485 (11) | 9.9202 (16) | 33.4862 (31) | 49.2842 (21) | 78.8995 (32)

16. Secondary Outcome: Part 2: Cmax,ss: Maximum Observed Plasma Concentration at Steady State for TAK-653
Time Frame: Day 18 pre-dose and at multiple time points (up to 24 hours) post dose
Population: The PK analysis set included all participants who received study drug and had at least 1 measurable plasma concentration or amount of drug in urine. The PK analysis population where data at specified time points was available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 2 Cohort 1: TAK-653 0.3 mg | Part 2 Cohort 2: TAK-653 1 mg | Part 2 Cohort 3: TAK-653 3 mg | Part 2 Cohort 4: TAK-653 6 mg | Part 2 Cohort 5: TAK-653 9 mg
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6
ng/mL | 7.6221 (29) | 23.9972 (31) | 97.2781 (28) | 140.4824 (37) | 223.3637 (53)

17. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-653 on Day 1
Time Frame: Part 1 Cohort 1-5: Day 1 pre-dose and at multiple timepoints (up to 144 hours) post-dose; Part 1 Cohort 6: Day 1 pre-dose and at multiple timepoints (up to 168 hours) post-dose; Part 2: Day 1 pre-dose and at multiple timepoints up to 120 hours) post-dose
Population: as for outcome 15
Measure: Median (Full Range); unit: hours
Arm/Group | Part 1 Cohort 1: TAK-653 0.3 mg | Part 1 Cohort 2: TAK-653 1 mg | Part 1 Cohort 3: TAK-653 3 mg+TAK-653 3mg | Part 1 Cohort 4: TAK-653 5 mg | Part 1 Cohort 5: TAK-653 9 mg | Part 1 Cohort 6: TAK-653 18 mg | Part 2 Cohort 1: TAK-653 0.3 mg | Part 2 Cohort 2: TAK-653 1 mg | Part 2 Cohort 3: TAK-653 3 mg | Part 2 Cohort 4: TAK-653 6 mg | Part 2 Cohort 5: TAK-653 9 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
hours | 1.250 [1.00 to 1.50] | 2.500 [1.00 to 3.00] | 1.750 [1.00 to 10.07] | 2.750 [1.00 to 12.10] | 5.500 [1.50 to 12.00] | 5.050 [1.00 to 10.03] | 1.250 [1.00 to 8.13] | 4.000 [1.00 to 6.00] | 1.500 [1.00 to 6.00] | 5.000 [3.00 to 6.08] | 4.508 [1.00 to 12.12]

18. Secondary Outcome: Part 2: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-653 on Day 18
Time Frame: Day 18 pre-dose and at multiple time points (up to 24 hours) post dose
Population: as for outcome 16
Measure: Median (Full Range); unit: hours
Arm/Group | Part 2 Cohort 1: TAK-653 0.3 mg | Part 2 Cohort 2: TAK-653 1 mg | Part 2 Cohort 3: TAK-653 3 mg | Part 2 Cohort 4: TAK-653 6 mg | Part 2 Cohort 5: TAK-653 9 mg
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6
hours | 2.500 [1.50 to 6.00] | 4.500 [2.00 to 12.00] | 4.000 [1.00 to 6.17] | 3.050 [1.00 to 10.00] | 3.000 [1.50 to 8.00]

19. Secondary Outcome: AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-653
Time Frame: as for outcome 17
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Part 1 Cohort 1: TAK-653 0.3 mg | Part 1 Cohort 2: TAK-653 1 mg | Part 1 Cohort 3: TAK-653 3 mg+TAK-653 3mg | Part 1 Cohort 4: TAK-653 5 mg | Part 1 Cohort 5: TAK-653 9 mg | Part 1 Cohort 6: TAK-653 18 mg | Part 2 Cohort 1: TAK-653 0.3 mg | Part 2 Cohort 2: TAK-653 1 mg | Part 2 Cohort 3: TAK-653 3 mg | Part 2 Cohort 4: TAK-653 6 mg | Part 2 Cohort 5: TAK-653 9 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
nanogram*hour per milliliter (ng*hr/mL) | 122.9927 (24) | 539.0930 (34) | 1310.5344 (23) | 2247.5468 (29) | 4264.3612 (37) | 7755.4570 (34) | 115.5869 (22) | 382.2871 (28) | 1417.0994 (31) | 1810.5437 (42) | 4065.9350 (54)

20. Secondary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-653
Time Frame: as for outcome 17
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Part 1 Cohort 1: TAK-653 0.3 mg | Part 1 Cohort 2: TAK-653 1 mg | Part 1 Cohort 3: TAK-653 3 mg+TAK-653 3mg | Part 1 Cohort 4: TAK-653 5 mg | Part 1 Cohort 5: TAK-653 9 mg | Part 1 Cohort 6: TAK-653 18 mg | Part 2 Cohort 1: TAK-653 0.3 mg | Part 2 Cohort 2: TAK-653 1 mg | Part 2 Cohort 3: TAK-653 3 mg | Part 2 Cohort 4: TAK-653 6 mg | Part 2 Cohort 5: TAK-653 9 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
ng*hr/mL | 143.6521 (29) | 596.5323 (43) | 1419.4306 (26) | 2536.8525 (35) | 4932.8519 (48) | 8413.1768 (40) | 129.5373 (26) | 448.9862 (36) | 1773.6365 (40) | 2027.7989 (56) | 5066.5536 (69)

21. Secondary Outcome: Part 2: AUCτ: Area Under the Plasma Concentration-time Curve From Time 0 to Time Tau Over the Dosing Interval for TAK-653
Time Frame: Days 6 and 18 pre-dose and at multiple timepoints (up to 24 hours) post-dose
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Part 2 Cohort 1: TAK-653 0.3 mg | Part 2 Cohort 2: TAK-653 1 mg | Part 2 Cohort 3: TAK-653 3 mg | Part 2 Cohort 4: TAK-653 6 mg | Part 2 Cohort 5: TAK-653 9 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
ng*hr/mL
  Day 6: number analyzed (Participants) | 6 | 6 | 6 | 5 | 6
  Day 6 | 51.0759 (19) | 159.9789 (16) | 578.9157 (26) | 778.2945 (13) | 1485.5059 (39)
  Day 18: number analyzed (Participants) | 6 | 6 | 6 | 5 | 6
  Day 18 | 144.7834 (32) | 477.3427 (38) | 1901.4065 (24) | 2747.5976 (42) | 4144.0176 (60)

22. Primary Outcome: Part 2: Number of Participants With Treatment-emergent Suicidal Ideation or Suicidal Behavior as Measured Using C-SSRS
Description: as for outcome 13
Time Frame: Baseline up to Day 21
Population: The safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Part 2 Cohorts 1-5: Pooled Placebo | Part 2 Cohort 1: TAK-653 0.3 mg | Part 2 Cohort 2: TAK-653 1 mg | Part 2 Cohort 3: TAK-653 3 mg | Part 2 Cohort 4: TAK-653 6 mg | Part 2 Cohort 5: TAK-653 9 mg
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
participants | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug up to Day 14 in Part 1 and Day 31 in Part 2
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Part 1 Cohorts 1-6: Pooled Placebo | Part 1 Cohort 1: TAK-653 0.3 mg | Part 1 Cohort 2: TAK-653 1 mg | Part 1 Cohort 3: TAK-653 3 mg+TAK-653 3mg | Part 1 Cohort 4: TAK-653 5 mg | Part 1 Cohort 5: TAK-653 9 mg | Part 1 Cohort 6: TAK-653 18 mg | Part 2 Cohorts 1-5: Pooled Placebo | Part 2 Cohort 1: TAK-653 0.3 mg | Part 2 Cohort 2: TAK-653 1 mg | Part 2 Cohort 3: TAK-653 3 mg | Part 2 Cohort 4: TAK-653 6 mg | Part 2 Cohort 5: TAK-653 9 mg
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/10 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/10 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 5/12 | 4/6 | 4/6 | 3/6 | 5/6 | 2/6 | 2/6 | 5/10 | 3/6 | 3/6 | 6/6 | 2/6 | 3/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 Cohorts 1-6: Pooled Placebo (N=12) | Part 1 Cohort 1: TAK-653 0.3 mg (N=6) | Part 1 Cohort 2: TAK-653 1 mg (N=6) | Part 1 Cohort 3: TAK-653 3 mg+TAK-653 3mg (N=6) | Part 1 Cohort 4: TAK-653 5 mg (N=6) | Part 1 Cohort 5: TAK-653 9 mg (N=6) | Part 1 Cohort 6: TAK-653 18 mg (N=6) | Part 2 Cohorts 1-5: Pooled Placebo (N=10) | Part 2 Cohort 1: TAK-653 0.3 mg (N=6) | Part 2 Cohort 2: TAK-653 1 mg (N=6) | Part 2 Cohort 3: TAK-653 3 mg (N=6) | Part 2 Cohort 4: TAK-653 6 mg (N=6) | Part 2 Cohort 5: TAK-653 9 mg (N=6)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Catheter site phlebitis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site related reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electroencephalogram abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 3 (4) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (3) | 2 (3) | 3 (5) | 1 (2) | 1 (2)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site discolouration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Puncture site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2017-03-24): https://cdn.clinicaltrials.gov/large-docs/56/NCT02561156/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-22): https://cdn.clinicaltrials.gov/large-docs/56/NCT02561156/SAP_001.pdf